CLINICAL TRIAL: NCT05978635
Title: Goal Directed Numeric Coaching as a Means of Preoxygenation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Thomas Jefferson University (Other)
Responsible Party: Principal Investigator, Stephen McNulty, Doctor of Osteopathic Medicine, Thomas Jefferson University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 16D.091
Record Dates: First submitted 2023-07-12; First posted 2023-08-07 (Actual); Last update posted 2023-08-07 (Actual); Status verified 2023-07

CONDITIONS: Pre-oxygenation
Keywords: Pre-oxygenation, vital capacity breaths

STUDY DESIGN:
Intervention Model Description: Once an adequate seal with consistent end tidal carbon dioxide on capnography is achieved, time starts. Patients are divided into two groups:
  Group A: Anesthesia provider encourages patient to breathe deeply by intermittently stating "take as deep a breath as you can". No goal directed numeric coaching is given. End point is 80% expired oxygen. The time it takes to achieve this end point and breath volumes are recorded.
  Group B: Anesthesia provider gives goal directed numeric coaching. For example, if the initial tidal volume achieved by the patient is 500mL, the provider states, "that was a 500mL breath, now try to achieve a 1000mL breath". The numeric goal should continue to increase above the patient's actual tidal volume (volume moved in and out of lungs during normal, quiet breathing) until an end point of 80% is reached. The time it takes to achieve this end point and breath volumes are recorded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Placebo Comparator): Anesthesia provider asks the patient to take 4 deep breaths by intermittently stating "take as deep a breath as you can". This is the standard of care technique for preoxygenation before induction of general anesthesia with the end point being 80% expired oxygen. The breath volumes in milliliters are recorded but not stated to the patient.
  Interventions: Behavioral: Group A Standard 4 deep breaths measured in milliliters from the ventilator.
- Group B (Experimental): Anesthesia provider asks the patient to take 4 deep breaths but provides coaching by informing the patient of the numeric volume (milliliters) to reach for every breath. Each tidal volume breath is measured using the anesthesia ventilator and the provider encourages the patient to achieve a higher tidal volume than previously achieved. For example, if the initial tidal volume achieved by the patient is 500 milliliter, the provider states, "that was a 500 milliliter breath, now try to achieve a 1000mL breath". The numeric goal should continue to increase above the patient's actual tidal volume. The breath volumes are recorded.
  Interventions: Behavioral: Group B Coached 4 deep breaths measured in milliliters from the ventilator

INTERVENTIONS:
Behavioral: Group A Standard 4 deep breaths measured in milliliters from the ventilator. — Tidal volume breath measured in milliliters
  Arms: Group A
Behavioral: Group B Coached 4 deep breaths measured in milliliters from the ventilator — Coached tidal volume breath measured in milliliters
  Arms: Group B

SUMMARY:
Pre-oxygenation is an anesthetic technique that allows for extended apneic (suspension of breathing) time prior to attempted endotracheal intubation. A common method to achieve adequate pre-oxygenation is having a patient take four vital capacity breaths of 100% oxygen in thirty seconds. This study seeks to determine if goal directed numeric coaching can lead to more accurate vital capacities during this technique.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists Physical Status 1 and 2
* nonsmokers
* primary English speaking
* undergoing elective surgery with planned endotracheal intubation

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2016-03-17 (Actual); Primary Completion 2018-12-20 (Actual); Study Completion 2018-12-20 (Actual)

PRIMARY OUTCOMES:
Vital capacity breaths measured in milliliters | Pre oxygenation period prior to induction of general anesthesia
  Measured vital capacity breaths volume in milliliters

IPD SHARING:
Plan to Share IPD: No